CLINICAL TRIAL: NCT00994669
Title: Development of a Non-invasive Assessment of Skeletal Muscle Loss in Cancer Patients
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 09-150B; 5R01CA127971 (NIH)
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Cachexia
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- healthy control male
- lung cancer male

SUMMARY:
The long-term objective of this research is to develop a non-invasive approach for early assessment of which patients are at high risk for future development of skeletal muscle atrophy. The investigators hypothesize that the rate constant for the terminal portion of the isotope decay curve following ingestion of a single oral dose of deuterated-3-methylhistidine (D-3MH) provides an accurate measure of this increased risk and that this rate constant can be measured non-invasively from timed spot urine samples. In addition, the investigators hypothesize that ingestion of a meat-containing meal will stimulate synthesis of skeletal muscle proteins to a greater extent than a non-meat-containing meal.

ELIGIBILITY:
Inclusion Criteria:

* male
* 30-85 years
* Body Mass Index (BMI) <30 kg/m2

Exclusion Criteria:

* Uncontrolled hypertension
* Glomerular filtration rate less than 60 mL/min/1.73 m2
* History of recurrent gastrointestinal bleeding
* Unable or unwilling to provide informed consent
* Ongoing anti-coagulant therapy

Ages: 30 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample of healthy males and male lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Assessment of the slope of terminal D-3MH/3MH decay curve post-dosing. | Post-dosing 12 to 22 hours
  Assess the slope of the terminal D-3MH/3MH decay curve for the post-dosing time period as calculated using plasma or urine samples and after a meat-containing or meat-free test meal.

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Sheffield-Moore, Ph.D., Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States